CLINICAL TRIAL: NCT05088265
Title: Prospective Real World Data Collection for the Bigfoot Unity Diabetes Management System
Brief Title: Bigfoot Unity Real World Study
Acronym: BURST
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Bigfoot Biomedical Inc. (Industry)
Collaborators: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Other Study IDs: 21BF01
Record Dates: First submitted 2021-10-08; First posted 2021-10-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Type 1 or Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Bigfoot Unity Diabetes Management System — The Bigfoot Unity System is a wirelessly connected set of hardware and software that is intended for use by people with diabetes mellitus who use disposable insulin pens for self-injection of insulin. Bigfoot Unity consists of the Abbott FreeStyle Libre 2 Sensor, two durable insulin pen caps (one each for specific rapid-acting and long-acting insulin pens) and an iOS-specific mobile App.

SUMMARY:
This study is observational, designed to collect real world use and safety data for those using the Bigfoot Unity Diabetes Management System for 12 months. Participants will be those with a prescription to use the Bigfoot Unity System. Medical practices prescribing Bigfoot Unity and Sponsor representatives will provide information about the study to current users and individuals considering initiation of the Bigfoot Unity System. During the course of the study, participants will be asked to use the Bigfoot Unity System in accordance with the prescription provided by their healthcare professional (HCP).

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 or type 2 diabetes diagnosis
2. HCP-prescribed, registered Bigfoot Unity users who have used the Bigfoot Unity System 2 weeks or less
3. Age 12 years or older at time of electronic informed consent
4. Using both long-acting and rapid-acting insulins that are compatible for use with the Bigfoot Unity System
5. Using long-acting insulin no more than 1 time per day
6. Must have baseline HbA1c collected within 90 days prior to starting the Bigfoot Unity System
7. Able to read and understand English
8. Participant or legally authorized representative for minors has the capacity to provide electronic informed consent
9. Resident of the United States
10. Persons who are using a phone that is compatible with Bigfoot Unity and not shared with a family member or a caregiver

Exclusion Criteria:

1. Females who are pregnant or intending to become pregnant during participation in the study
2. Persons with implantable medical devices such as pacemakers
3. Persons on dialysis or other serious medical conditions that would impact the ability to use the device or manage their diabetes
4. Persons taking or expected to be taking >500mg Vitamin C supplements on routine basis
5. Persons employed by the Sponsor or JCHR

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of users 12 years or older who have type 1 or type 2 diabetes who are prescribed the Bigfoot Unity Diabetes Management System for managing their diabetes for multiple daily injections consistent with the labeling of the product.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-10-26 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | 3 months
  Glycated hemoglobin
Change from baseline in HbA1c | 6 months
  Glycated hemoglobin
Change from baseline in HbA1c | 9 months
  Glycated hemoglobin
Change from baseline in HbA1c | 12 months
  Glycated hemoglobin
Percent time Sensor in range of 70 mg/dL to 180 mg/dL, inclusive | 3 months
Percent time Sensor in range of 70 mg/dL to 180 mg/dL, inclusive | 6 months
Percent time Sensor in range of 70 mg/dL to 180 mg/dL, inclusive | 9 months
Percent time Sensor in range of 70 mg/dL to 180 mg/dL, inclusive | 12 months
Glucose management indicator | 3 months
Glucose management indicator | 6 months
Glucose management indicator | 9 months
Glucose management indicator | 12 months
Percent time Sensor in hypoglycemia | 3 months
  Will evaluate Sensor below 70 mg/dL and below 54 mg/dL
Percent time Sensor in hypoglycemia | 6 months
  Will evaluate Sensor below 70 mg/dL and below 54 mg/dL
Percent time Sensor in hypoglycemia | 9 months
  Will evaluate Sensor below 70 mg/dL and below 54 mg/dL
Percent time Sensor in hypoglycemia | 12 months
  Will evaluate Sensor below 70 mg/dL and below 54 mg/dL
Percent time Sensor in hyperglycemia | 3 months
  Will evaluate Sensor above 180 mg/dL and above 250 mg/dL
Percent time Sensor in hyperglycemia | 6 months
  Will evaluate Sensor above 180 mg/dL and above 250 mg/dL
Percent time Sensor in hyperglycemia | 9 months
  Will evaluate Sensor above 180 mg/dL and above 250 mg/dL
Percent time Sensor in hyperglycemia | 12 months
  Will evaluate Sensor above 180 mg/dL and above 250 mg/dL
Change from baseline in Diabetes Distress Scale | 3 months
  Measures emotional and behavioral challenges generated by diabetes and its management; scale is 1.0 to 6.0, higher scores are worse.
Change from baseline in Diabetes Distress Scale | 6 months
  Measures emotional and behavioral challenges generated by diabetes and its management; scale is 1.0 to 6.0, higher scores are worse.
Change from baseline in Diabetes Distress Scale | 9 months
  Measures emotional and behavioral challenges generated by diabetes and its management; scale is 1.0 to 6.0, higher scores are worse.
Change from baseline in Diabetes Distress Scale | 12 months
  Measures emotional and behavioral challenges generated by diabetes and its management; scale is 1.0 to 6.0, higher scores are worse.
Change from baseline in Hypoglycemia Confidence Scale | 3 months
  Measures the degree to which people with diabetes feel able, secure, and comfortable regarding their ability to stay safe from hypoglycemic-related problems; scale is 1.0 to 4.0, higher scores are worse.
Change from baseline in Hypoglycemia Confidence Scale | 6 months
  Measures the degree to which people with diabetes feel able, secure, and comfortable regarding their ability to stay safe from hypoglycemic-related problems; scale is 1.0 to 4.0, higher scores are worse.
Change from baseline in Hypoglycemia Confidence Scale | 9 months
  Measures the degree to which people with diabetes feel able, secure, and comfortable regarding their ability to stay safe from hypoglycemic-related problems; scale is 1.0 to 4.0, higher scores are worse.
Change from baseline in Hypoglycemia Confidence Scale | 12 months
  Measures the degree to which people with diabetes feel able, secure, and comfortable regarding their ability to stay safe from hypoglycemic-related problems; scale is 1.0 to 4.0, higher scores are worse.
Change from baseline in Insulin Delivery Satisfaction Survey | 3 months
  Measures the effectiveness, burdensomeness and inconvenience of an insulin delivery system; scale is 1.0 to 5.0, higher scores are better.
Change from baseline in Insulin Delivery Satisfaction Survey | 6 months
  Measures the effectiveness, burdensomeness and inconvenience of an insulin delivery system; scale is 1.0 to 5.0, higher scores are better.
Change from baseline in Insulin Delivery Satisfaction Survey | 9 months
  Measures the effectiveness, burdensomeness and inconvenience of an insulin delivery system; scale is 1.0 to 5.0, higher scores are better.
Change from baseline in Insulin Delivery Satisfaction Survey | 12 months
  Measures the effectiveness, burdensomeness and inconvenience of an insulin delivery system; scale is 1.0 to 5.0, higher scores are better.
System Usability Scale | 3 months
  Measures the usability of a system; scale is 0 to 100, higher scores are better.
System Usability Scale | 6 months
  Measures the usability of a system; scale is 0 to 100, higher scores are better.
System Usability Scale | 9 months
  Measures the usability of a system; scale is 0 to 100, higher scores are better.
System Usability Scale | 12 months
  Measures the usability of a system; scale is 0 to 100, higher scores are better.

CONTACTS AND LOCATIONS:
Overall Officials: Jim Malone, MD, Principal Investigator — Bigfoot Biomedical
Locations (1):
- Bigfoot Biomedical Inc., Milpitas, California, United States

IPD SHARING:
Plan to Share IPD: No